| AtaCor Medical, Inc. | | | Revision A |
|---|---|---|---|
| Clinical Investi | igation Plan Synopsis - Subcostal Temporary Extracardiac Pacing (S | TEP) Study | |
| Excerpt of DOC-10052 | | | |



## **Synopis of Clinical Investigation Plan (CIP)**

Subcostal Temporary Extracardiac Pacing (STEP) Study

Clinical Study of the AtaCor Extracardiac Pacing System

Excerpt from DOC-10052, Revision A

23 July, 2019

NCT 04096365

## **SPONSOR:**

ATACOR MEDICAL, INC.
635 CAMINO DE LOS MARES, SUITE 205
SAN CLEMENTE, CA 92673

| AtaCor Medical, Inc. | ] | Revision A |
|---|---|---|
| Clinical Investigation Plan Synopsis – Subcostal Temporary Extracardiac Pacing (STEP) Study | | |
| Excerpt of DOC-10052 | ] | |

## **Synopsis of the Clinical Investigation**

| Study Name | Subcostal Temporary Extracardiac Pacing (STEP) Study |
|---|---|
| Study<br>Objectives | To evaluate initial safety and performance of the AtaCor Temporary Pacing System. Safety will be evaluated through analysis of all Adverse Events. Performance will be evaluated through (1) the incidence of successful StealthTrac Lead placement using the MACH I Delivery Tool, (2) measurements of capture thresholds, sensed R-wave amplitudes, pacing impedance and concomitant skeletal muscle stimulation at rest, in multiple postures and during in-hospital ambulation, and (3) differences in cardiac conduction (12 lead ECG) and function (Echocardiography) while pacing with temporary transvenous lead, the AtaCor StealthTrac Lead and during intrinsic conduction. |
| Study Size | Up to 15 Subjects inserted with the StealthTrac Lead from a maximum of three (3) investigation sites. This study is not statistically-powered. Results may be used to generate hypotheses for subsequent clinical investigations. |
| Study<br>Duration | The total expected duration of the investigation is four (4) to six (6) months, comprising two (2) to four (4) months for enrollment and follow-up, plus an additional two (2) months to analyze study data and prepare a final report. Subject participation consists of an in-hospital device evaluation up to seven (7) days and a 30-day post-removal follow-up visit to detect any latent adverse events after hospital discharge. |
| Study Design | Prospective, subacute (in-hospital), single-arm, multicenter |
| Study<br>Population | <ol> <li>To participate in this clinical investigation, Subjects must meet all the following criteria: <ol> <li>Indicated for closed-chest cardiac invasive procedure with the potential for intra-procedural or post-procedural bradycardia and willing to be hospitalized for a minimum of 2 days post procedure.</li></ol></li></ol> |

| AtaCor Medical, Inc. | | Revision A |
|---|---|---|
| Clinical Invest | igation Plan Synopsis - Subcostal Temporary Extracardiac Pacing (STEP) Study | |
| Excerpt of DOC-10052 | | |

Figure 1 provides an Eligibility Criteria Met + Written Informed Consent overview of study **Enrollment** Demographics, Medical History & Medications Review activities. Enrolled Subjects will have a Insert Market Released & StealthTrac Pacing Leads market-released Electrical Performance Evaluations (both leads) transvenous pacing lead Pre-/Post-StealthTrac implant echo for PE investigational and Index Procedure (e.g. TAVR, BAV, PPM) StealthTrac Lead placed. **Index Visit** Final Electrical Performance Evaluation (both leads) Both leads will be Evaluate High Rate Pacing with StealthTrac Pacing Lead evaluated to confirm X-ray to document lead positions ventricular sensing and capture. Diagnostic echocardiograms will be Market Released Lead Electrical Performance performed to detect any Evaluation (single posture) pericardial effusions StealthTrac Electrical Performance Evaluation (multiple caused by inserting the postures) StealthTrac Lead. The 12 Lead ECG and Subject Perception Questionnaire index procedure will be during pacing with both leads **In-Hospital** performed according to Investigator interview for usability and human factors standard of care Stay Holter evaluation and patient questionnaire regarding methods, after which the (2 to X days; discomfort and mobility restrictions StealthTrac Lead will be Final X-Ray to document lead position prior to removal up to 7) used to deliver high rate of the StealthTrac Lead pacing (160 to 220 Final echo for latent PE and cardiac function BPM) in clinically Market Released Lead removal appropriate Subjects. StealthTrac Lead removal prior to discharge (pre-The electrical removal x-ray for lead position) performance of both Patient questionnaire regarding removal leads will be reconfirmed, and lead **Final** positions will he 30-day post-removal follow-up to detect any latent AEs Follow-up documented using x-ray before the Subject leaves the procedure room. The Figure 1. Study Flow Chart day after the procedure,

Subjects will undergo a 12 lead ECG while pacing with each lead.

Both leads will undergo daily Electrical Performance Evaluations and in multiple postures when clinically appropriate. Post-operative evaluations will be performed during periods of rest and during activity. Appropriate pacing performance during activity will be evaluated using ECG Holter monitor recordings. Subjects will also be asked patient-centric questions about their experience with the StealthTrac Lead throughout the study period.

Evaluations will continue until the Subject is discharged from the hospital, with a minimum of two (2) and a maximum of seven (7) evaluation days after the index procedure. Prior to StealthTrac Lead removal, an X-Ray will be taken to document the final lead position and diagnostic echocardiography will be performed to (1) detect any latent pericardial effusions and (2) assess differences in cardiac function with intrinsic conduction and while pacing with the StealthTrac Lead and market released lead. A final follow-up will be performed 25-30 days after removal to identify any latent adverse events before the Subject exits the study.